CLINICAL TRIAL: NCT03209453
Title: Therapeutic Effects of Short-term Family-centered Work Shop for Children With Developmental Delays: a Randomized Trial
Brief Title: Effects of Family Work Shop for Children With Developmental Delays: a Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DOH-SKH-106
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Development Delay
Keywords: family work shop
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): children with developmental delays, under regular rehabilitation programs, participate the family work shop family work shop: 6 families in one course, 2 hours per session, one session per week, a total of 6 weeks
  Interventions: Other: family work shop
- control group (No Intervention): children with developmental delays, under regular rehabilitation programs, not participate the family work shop

INTERVENTIONS:
Other: family work shop — Children with developmental delays, under regular rehabilitation programs, participate 6 sessions of family work shop The family work shop had 6 families in one course, 2 hours per week, for a total of 6 weeks.
  Arms: study group

SUMMARY:
To identify the therapeutic effects of short-term family-centered work shop for children with developmental delays

DETAILED DESCRIPTION:
1. The family work shop has a total of 6 weeks, with 6 families in one course. 2. Two hours per session, one time per week. Aims;

1. Assess the effects of family work shop for children with developmental delays, including functional performance and health-related quality of life.
2. Assess the family strain by work shop for parents of children with developmental delays.

ELIGIBILITY:
Inclusion Criteria:

* 18 M/O to 36 M/O children with developmental delays, under regular rehabilitation programs

Exclusion Criteria:

* less than 18 M/O and older than 36 M/O failed to obtain written informed consent

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline functional performance (scores) at 6 weeks | baseline and up to 6 weeks
  Pediatric Outcome Data Collection Instrument

SECONDARY OUTCOMES:
change from baseline health-related quality of life (scores) at 6 weeks | baseline and up to 6 weeks
  Child Health Questionnaire
change from baseline caregiver health-related quality of life (scores) at 6 weeks | baseline and up to 6 weeks
  World Health Organization Quality of Life: brief form
change from baseline family strain (scores) at 6 weeks | baseline and up to 6 weeks
  Caregiver strain index
change from baseline family impact | baseline and up to 6 weeks
  Pediatric Quality of Life Inventory: Family impact module

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No